CLINICAL TRIAL: NCT05640778
Title: Efficacy and Safety of Neoadjuvant Dalpiciclib Combined With Endocrine Therapy in Luminal B/HER2-negative Breast Cancer and Biomarker Analysis: a Single-arm, Open-label Trial
Brief Title: Neoadjuvant Dalpiciclib Plus Aromatase Inhibitors in Luminal B/HER2-negative Breast Cancer (DANCER)
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Collaborators: GeneCast Biotechnology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2022-0500
Record Dates: First submitted 2022-11-30; First posted 2022-12-07 (Actual); Last update posted 2024-01-31 (Actual); Status verified 2023-10

CONDITIONS: Luminal B/HER2-negative Breast Cancer
MeSH Terms: interventions — Aromatase Inhibitors

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- neoadjuvant endocrine therapy (Experimental): CDK4/6 inhibitor combined with aromatase inhibitor
  Interventions: Drug: Dalpiciclib combined with aromatase inhibitors

INTERVENTIONS:
Drug: Dalpiciclib combined with aromatase inhibitors — Dalpiciclib combined with letrozole or anastrozole

SUMMARY:
Evaluate the efficacy and safety of Dalpiciclib combined with aromatase inhibitors as a neoadjuvant therapy in Luminal B/HER2-negative breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Patient is ≥ 18 years-old at the time of consent to participate this trial
* Famale stage I-III breast cancer patients
* HR-positive（ER≥10%）, HER2-negtive invasive breast cancer, either Ki67≥20% and/or PgR<20%
* No prior anti-cancer treatment
* ECOG 0-1

Exclusion Criteria:

* Known to have other aggressive malignant tumor in the past 5 years.
* Bilateral breast cancer; Inflammatory breast cancer; Occult breast cancer; Distant metastasis confirmed by pathology.
* There are other concomitant diseases that seriously threaten the patient's safety or affect the patient's completion of the study, such as serious infection, liver disease, cardiovascular disease, kidney disease, respiratory disease or uncontrolled diabetes or dyslipidemia.
* Female patients during pregnancy or lactation.
* The investigator determines that subjects are not appropriate to participate in the study due to other factors.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-10-01 (Actual); Primary Completion 2024-10-31 (Estimated); Study Completion 2025-10-31 (Estimated)

PRIMARY OUTCOMES:
Complete cell cycle arrest（CCCA, defined as ki67≤2.7%）rate at 2 weeks of treatment | 3 years
  Assess ki67 level through biopsy samples of patients

SECONDARY OUTCOMES:
Objective response rate (ORR) | 3 years
  the proportion of people with clinical complete response(CR) or partial response(PR), per RECIST v1.1

CONTACTS AND LOCATIONS:
Locations (1):
- 2nd Affiliated Hospital, School of Medicine, Zhejiang University, Hangzhou, China

IPD SHARING:
Plan to Share IPD: Undecided